CLINICAL TRIAL: NCT01894711
Title: Real-world Use and (Cost)-Effectiveness of Adjuvant Trastuzumab in Early Breast Cancer
Brief Title: Real World Efficiency of Trastuzumab in Early Breast Cancer
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MEC 09-4-075
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with HER2 positive tumors: Patients with HER2 positive tumors treated with trastuzumab or not treated with trastuzumab
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Treatment with trastuzumab in HER2 positive patients
  Other Names: Herceptin

SUMMARY:
AIM To determine the value of trastuzumab in the early breast cancer setting in the Netherlands.

RESEARCH QUESTIONS / OBJECTIVES

1. Is adjuvant trastuzumab in daily practice effectively used, that is, how and to whom is it given?
2. Is the introduction of trastuzumab in early breast cancer cost-effective for the Netherlands?

To address the research questions (objectives), the following outcome measures will be determined:

CLINICAL OUTCOME MEASURES

1. Actual trastuzumab administration as opposed to planned trastuzumab administration
2. Selection criteria for chemotherapy and trastuzumab in daily practice
3. Immediate and longterm toxicities due to adjuvant treatment, specifically cardiac
4. Disease-free, breast cancer specific, and overall survival in relation to trastuzumab

   ECONOMIC OUTCOME MEASURES
5. Volumes and costs of diagnostic tests and therapies including those for (distant) relapse
6. Cost-effectiveness of trastuzumab in clinical trials versus in real world

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with invasive stage I-III breast cancer in the years 2005, 2006 and 2007 in the participating 5 hospitals.

Exclusion Criteria:

* Distant metastasis at the time of the primary diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with invasive stage I-III breast cancer in the years 2005, 2006 and 2007 in the participating 5 hospitals.
  That is, no distant metastasis at the time of the primary diagnosis
Sampling Method: Probability Sample
Enrollment: 2684 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the use of trastuzumab in patients with human epidermal growth factor receptor 2 (HER2) positive tumor | events, within an average of 5-year between diagnosis and last follow up
  Disease free survival

SECONDARY OUTCOMES:
Number of patients treated with trastuzumab who develop (cardio)toxicity? | temporary or definite stop trastuzumab, within an average of 5-year between diagnosis and last follow up
  cardiotoxicity

OTHER OUTCOMES:
Cost-effectiveness os trastuzumab in adjuvant breast cancer patients | volume and cost, within an average of 5-year between diagnosis and last follow up

CONTACTS AND LOCATIONS:
Overall Officials: Vivianne CG Tjan-Heijnen, MD., Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands